CLINICAL TRIAL: NCT05892237
Title: Bronchial Artery Interventional Therapy and Sequential Radiotherapy in the Treatment of Non-resectable, Non-metastatic Central-type Squamous Lung Cancer
Brief Title: CIETAI and Sequential Radiotherapy in Squamous Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dong Wang (Other)
Responsible Party: Sponsor-Investigator, Dong Wang, dean of clinical oncology (fomer), Third Military Medical University
Organization: Third Military Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023108
Record Dates: First submitted 2023-05-19; First posted 2023-06-07 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immunotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- central-type squamous NSCLC (Experimental): 1. Phase I:
  1. Chemo-Immulo-embolization via Tumor Arterial, CIETAI:
     DSA guided tumor artery infusion of nano-paclitaxel 200 mg+PD-1 inhibitor (Tirelizumab) 200mg, followed by gelatin sponge particles (350-560um) embolization
  2. two cycles of chemotherapy combined with immune checkpoint inhibitors (q3w): Nano-paclitaxel 260 mg/m2, d1, ivgtt; Cisplatin 75mg/m2, d1, ivgtt; PD-1 inhibitor (Tirelizumab) 200mg, d1, ivgtt, 30-60min 2. phase II: Chest radiotherapy: 60Gy/2Gy/30f 3. phase III: PD-1 inhibitor (Tirelizumab) 200mg, d1, ivgtt, 30-60min Maintenance for 1 year
  Interventions: Procedure: bronchial artery interventional therapy; Drug: Chemotherapy drug; Radiation: IMRT; Drug: Immunotherapy

INTERVENTIONS:
Procedure: bronchial artery interventional therapy — After successful anesthesia, right femoral artery puncture was performed by Seldinger method. 5F-Yashrio catheter is chosen to locate the bronchial artery of the diseased side at the level of the thoracic aortotracheal bifurcation. Angiography was performed (Osu 300mg/ml, 3ml/s, total 8ml, 200Psi) to visualize tumor blood supply artery before infusion of chemo+PD-1 inhibitor and embolism.
Drug: Chemotherapy drug — Nano-paclitaxel 260 mg/m2, d1, ivgtt, q3w+Cisplatin 75mg/m2, d1, ivgtt,q3w.
Radiation: IMRT — 60Gy/2Gy/30f
Drug: Immunotherapy — PD-1 inhibitor (Tirelizumab) 200mg, d1, ivgtt, 30-60min, q3w.

SUMMARY:
Central-type lung cancer refers to lung malignancies originating from the segmental bronchi and above. The most common tissue type is squamous cell carcinoma. Patients often present with cough, hemoptysis, hoarseness and also some critical conditions including superior vena caval obstruction syndrome. Therefore, effective treatment should be implemented as early as possible to rapidly reduce tumor burden and control the progression of the disease. Most of the central-type NSCLC are classified into T3-4, N1-2 stage and are non-resectable. The PACIFIC study changed the standard treatment model for inoperable locally advanced lung cancer with synchronous chemoradiotherapy and sequential PD-L1 immunotherapy. In clinical practice, Chinese patients often failed to finish concurrent chemoradiotherapy for high toxicity. In addition, combination with PD-1/PD-L1 inhibitors increased the risk of immune related pneumonia.

Bronchial artery infusion (BAI), that directly infused drugs (chemo and PD-1 inhibitor) through tumor-nourishing arteries, has potential advantages in the treatment of central-type lung cancer. The drug concentration in tumor region increased to potentiate the antitumoral effect and also reduced the systemic adverse reactions.

In this study, bronchial artery interventional therapy is conducted with precedence. The protocol for bronchial artery intervention includes infusion of chemo and PD-1 inhibitor followed by bronchial artery embolism (Chemo-Immulo-embolization via Tumor arterial, CIETAI). Followed CIETAI, two cycles of chemo/PD-1 therapy are planned to carried out before radiotherapy. After radiotherapy, maintenance PD-1 inhibitor are initiated for 1 year or until progression.

DETAILED DESCRIPTION:
PD-1/PD-L1 immune checkpoint inhibitor (ICI), which has been introduced in the treatment of lung cancer, gastric cancer, colorectal cancer and other solid tumors, changed the strategy of cancer treatment. The more widely biomarkers for its efficacy include tumor PD-L1 proportional score (TPS), tumor mutation burden (TMB), DNA mismatch repair defect (dMMR), genomic instability (MSI-H) which were used to assess PD-L1 expression in tumor cells and the presence and density of T cells in the tumor microenvironment (TME). However, the overall efficacy of PD-1/PD-L1 remain unsatisfactory. To increase the concentration of PD-1/PD-L1 inhibitor in tumor and TME is a potential strategy to increase the efficacy. In this study, perfusion of PD-1/PD-L1 via bronchial arterial was harnessed to maximize the concentration of drugs in the tumor. We proposed a surgical procedure called Chemo-Immuno-embolization via Tumor Arterial Intervention (CIETAI). This study mainly included inoperable patients with central-type lung squamous cell carcinoma who received CIETAI at the initial treatment, followed by radiotherapy and PD-1/PD-L1 maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Patients volunteered to participate in the study and signed the informed consent.
* Age 18-80, both male and female.
* Histologically or cytologically confirmed squamous lung cancer staging T3-4, Nany, and M0 (according to the American Joint Committee on Cancer Staging (AJCC) 2017 Edition 8 TNM Staging System). Central-type classified according to chest imaging or bronchoscopy.
* At least one measurable lesion according to RECIST 1.1.
* ECOG PS 0-1.
* Expected survival ≥ 6 months.
* Patients who never received systemic therapy in the past, including radiotherapy, chemotherapy, targeted therapy and immunotherapy, or patients who relapsed more than 6 months after adjuvant chemotherapy.
* The main organ functions accorded with the following criteria within 7 days before treatment:

  1. Blood routine examination ( without blood transfusion in 14 days): hemoglobin (HB) ≥ 90 g/L; neutrophil absolute value (ANC) ≥ 1.5 *109/L; platelet (PLT) ≥80 *109/L.
  2. Biochemical tests should meet the following criteria: 1) total bilirubin (TBIL) ≤1.5 times of upper limit of normal (ULN); 2) alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 *ULN, if accompanied by liver metastasis, ALT and AST ≤ 5* ULN; 3) serum creatinine (Cr) ≤ 1.5* ULN or creatinine clearance rate (CCr) ≥ 60 ml/min;4) Serum albumin (≥35g/L). (3) Doppler echocardiography: left ventricular ejection fraction (LVEF) ≥the low limit of normal value (50%).
* Tissue samples should be provided for biomarker analysis (such as PD-L1) Patients who could not provide new tissues could provide 5-8 paraffin sections of 3-5 μm by archival preservation. Blood sample should be collected at a pre-specified time point to complete the continuous dynamic MRD analysis. (non-mandatory).

Exclusion Criteria:

* Severe allergic reactions to humanized antibodies or fusion proteins in the past.
* Severe allergic reactions to component contained in contrast agent or granule embolism agent in the past.
* Metastasis to bone, brain, liver, pleural cavity, or any other distant organs.
* Diagnosed of immunodeficiency or received systemic glucocorticoid therapy or any other form of immunosuppressive therapy within 14 days before the study, allowing physiological doses of glucocorticoids (≤10mg/day prednisone or equivalent).
* Patients with active, known or suspected autoimmune diseases. Patients with type I diabetes, hypothyroidism requiring hormone replacement therapy, skin disorders requiring no systemic treatment (such as vitiligo, psoriasis or alopecia). Patients who would not triggers can be included.
* Serious heart disease, include congestive heart failure, uncontrollable high-risk arrhythmia, unstable angina pectoris, myocardial infarction, and severe valvular disease.
* Patients received systemic antineoplastic therapy, including cytotoxic therapy, signal transduction inhibitors, immunotherapy (or mitomycin C within 6 weeks before the grouping),recieved over-extended-field radiotherapy (EF-RT) within 4 weeks before the grouping or limited-field radiotherapy to evaluate the tumor lesions within 2 weeks before the grouping.
* Positive hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus antibody (HCV Ab), indicating acute or chronic infection.
* Patients with active pulmonary tuberculosis (TB) infection judged by chest X-ray examination, sputum examination and clinical physical examination. Patients with active pulmonary tuberculosis infection in the previous year should be excluded even if they have been treated; Patients with active pulmonary tuberculosis infection more than a year ago should also be excluded unless the course and type of antituberculosis treatment previously were appropriate.
* Patients with brain metastases with symptoms or symptoms controlling less than 2 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate 2 (ORR2) | 2 year
  complete response(CR)+partial response(PR) according to RECIST 1.1

SECONDARY OUTCOMES:
Objective Response Rate 1 (ORR1) | 1 year
  complete response(CR)+partial response(PR) according to RECIST 1.1
Improvements of main symptoms after CITAI | 1 year
  NSCLC related symptoms evaluated by NSCLC-SAQ v1.0
Progression-free Survival(PFS) | approximately 10 months
  progression-free survival is defined as the time from enrollment to the date of first document disease progression or death from any cause
Overall Survival（OS) | approximately 18 months
  overall survival is defined as the time from randomization to death from any cause
Toxicity | the first date of treatment to 30 days after the last dose of study drug
  Summary of the adverse events experienced by study participants as evaluated by Common Terminology Criteria for Adverse Events (CTCAE) v5.0
EORTC QLQ-C30 | the first date of treatment to 30 days after the last dose of study drug
  according to EORTC QLQ-C30
EORTC QLQ-LC13 | the first date of treatment to 30 days after the last dose of study drug
  according to EORTC QLQ-LC13

OTHER OUTCOMES:
Tumor proportion score (TPS) of PD-L1 | Baseline
  IHC by 22C3 antibody
ctDNA MRD | Baseline and 30 days after the last dose of study drug
  ctDNA MRD detection by liquid biopsy change during treatment
Surgery rate | 2 year
  MDT to discuss surgery after phase I treatment and phase II treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No